CLINICAL TRIAL: NCT02916524
Title: Double-blind Randomized Trial Investigating the Use of Computational Modeling to Predict Rehabilitation Outcomes in Bilingual Aphasia
Brief Title: Predicting Rehabilitation Outcomes in Bilingual Aphasia Using Computational Modeling
Acronym: PROCoM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Boston University Charles River Campus (Other)
Collaborators: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Principal Investigator, Swathi Kiran, Professor, Boston University Charles River Campus
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 4492E; U01DC014922-01A1 (NIH)
Record Dates: First submitted 2016-09-16; First posted 2016-09-27 (Estimated); Last update posted 2021-04-19 (Actual); Status verified 2021-04

CONDITIONS: Aphasia
Keywords: Aphasia; Bilingualism; Language therapy; Rehabilitation of speech and language disorders; Speech-language pathology
MeSH Terms: conditions — Aphasia; Language Disorders

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Model-based (Experimental): Semantic Feature Analysis training will be provided in the language that was selected by the computational model.
  Interventions: Behavioral: Semantic Feature Analysis (SFA)
- Model-opposite (Active Comparator): Semantic Feature Analysis training will be provided in the language opposite to that which was selected by the computational model.
  Interventions: Behavioral: Semantic Feature Analysis (SFA)
- Sub-Study: Computational Modeling for Bilingual Dementia and Semantic Decline (No Intervention): This is a sub-study aimed at building a computational model to simulate bilingual dementia and semantic decline.

INTERVENTIONS:
Behavioral: Semantic Feature Analysis (SFA) — SFA training entails having the speech-language pathologist (SLP) guide the participant through generation of pertinent semantic features for pictured treatment items (e.g., category membership, physical description, location of item in context, action associated with item). Treatment is applied to a set of items in the context of single-subject, multiple baseline designs so that replication of treatment effects could be evaluated within and across participants. Treatment will be administered two times per week until prescribed accuracy levels were met during treatment probes or a maximum number of treatment sessions was completed.
  Arms: Model-based; Model-opposite

SUMMARY:
The purpose of this investigation is to implement a computational model that can predict and optimize training and cross-language generalization patterns for bilingual persons with aphasia (BPA). The proposed work will determine the best possible treatment program for each individual patient even before they are rehabilitated. In addition, the computational model allows specification of variables such as age of acquisition, language exposure/proficiency, impairment and their systematic influence on a range of language rehabilitation outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Any number of years of education
* Bilingual: speaking both Spanish and English (or Chinese and English) with any degree of language proficiency prior to stroke
* Aphasia secondary to a left-hemisphere stroke (diagnosed by a neurologist on the basis of clinical CT/MRI imaging or medical reports)
* Aphasia resulting from stroke or dementia
* Naming deficits must be present with concurrent lexical/semantic impairment
* Visual and auditory acuity sufficient for all assessment and treatment procedures
* Ability to understand study and follow study procedures for the entire length of the study

Exclusion Criteria:

* Premorbid history of speech/language disorder
* Proficient in more than just Spanish and English (or Chinese and English)
* Overt, behaviorally noticeable, attentional limitations that interfere with completing the experimental tasks
* Active medical disease that may compromise participation (e.g., cancer undergoing acute treatment, unstable diabetes, renal or hepatic insufficiency, fluctuating systemic immunological disease such as systemic lupus erythematosis, etc.)
* Currently taking medications that are known to exert significant effects on cognitive processes, such as neuroleptics, steroids, anticholinesterase inhibitors, etc.
* Current drug or alcohol use or dependence that would interfere with adherence to study requirements, in the opinion of the principal investigator
* Inability or unwillingness of individual to give written informed consent
* Diagnosed with mental illness other than active depression
* Neurological condition other than that which resulted in aphasia

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2018-04-20 (Actual); Primary Completion 2021-07-31 (Estimated); Study Completion 2023-07-31 (Estimated)

PRIMARY OUTCOMES:
Word Retrieval Accuracy in both languages | Through study completion, an average of 10 weeks
  Accuracy of naming of pictured treated and untreated items in both languages will be assessed in probes conducted separate from treatment. Probes were conducted repeatedly throughout the study, from baseline (prior to treatment) to the end of treatment. All naming responses were scored using as correct or incorrect. A percentage accuracy was calculated for each set of items for every probe session. Baseline probe scores were compared to end of treatment probe scores to obtain individual effect sizes for each sets of items for each participant (i.e., several effect sizes were calculated for each participant).

SECONDARY OUTCOMES:
Psycholinguistic assessments of language processing in aphasia (PALPA) in both languages | Week 1 and up to 10 weeks
  Reading single words and understanding spoken words
Boston Naming Test (BNT) in both languages | Week 1 and up to 10 weeks
  Naming pictured items
Bilingual Aphasia Test (BAT) B and C in both languages | Week 1 and up to 10 weeks
  Assesses each of the languages of a bilingual or multilingual individual with aphasia
Western Aphasia Battery (WAB) in both languages | Week 1 and up to 10 weeks
  Assesses the levels of impairment of aphasia
Cognitive Linguistic Quick Test (CLQT) in both languages | Week 1 and up to 10 weeks
  Assesses the contribution of cognitive deficits to language dysfunction
Verbal fluency task (COWAT) in both languages | Week 1 and up to 10 weeks
  Assesses general fluency
Category fluency task in both languages | Week 1 and up to 10 weeks
  Assesses category fluency
Communication Effectiveness Index (CETI) for both languages | Week 1 and up to 10 weeks
  Determines communication effectiveness by proxy
Pyramids and Palm Trees Test (PAPT) 3 pictures version | Week 1 and up to 10 weeks
  Assesses semantic processing ability
Aphasia Bank | Week 1 and up to 10 weeks
  Assesses discourse

CONTACTS AND LOCATIONS:
Overall Officials: Swathi Kiran, PhD, Principal Investigator — Boston University
Locations (3):
- United States (3):
  - San Francisco State University, San Francisco, California
  - Boston University Sargent College, Boston, Massachusetts
  - Austin Speech Labs, Austin, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Russell-Meill M, Carpenter E, Marte MJ, Scimeca M, Penaloza C, Kiran S. Measurement of cross-language and cross-domain generalization following semantic feature-based anomia treatment in bilingual aphasia. Neuropsychol Rehabil. 2025 Jun 26:1-27. doi: 10.1080/09602011.2025.2522196. Online ahead of print. PMID 40571559
- [Derived] Penaloza C, Dekhtyar M, Scimeca M, Carpenter E, Mukadam N, Kiran S. Predicting treatment outcomes for bilinguals with aphasia using computational modeling: Study protocol for the PROCoM randomised controlled trial. BMJ Open. 2020 Nov 18;10(11):e040495. doi: 10.1136/bmjopen-2020-040495. PMID 33208330
- See also: Aphasia Research Laboratory website — http://www.bu.edu/aphasiaresearch/